

| Official Title: | Impact of Online Ordering on Low-Income Adults' Food Security in Online Food Pantry Settings |
|---|---|
| NCT Number: | NCT05752721 |
| Study Number: | 22-01523 |
| Document Type: | Informed Consent Form |
| Date of the Document: | • May 9, 2023 |

Intervention Arm 



# Research Subject Consent/ Study Information Sheet

Title of Study: Impact of Online Ordering on Low-Income Adults' Food Security in Online Food

Pantry Settings s22-01523

**Principal** Pasquale Rummo, PhD **Investigator:** NYU Langone Health

Department of Population Health

180 Madison Avenue, 3rd floor, New York, New York 10016

Pasquale.Rummo@nyulangone.org

646-501-3371

**Emergency Contact:** Pasquale Rummo

646-501-3371

## 1. Key Study Information

You are being invited to take part in a research study. Participation is completely voluntary. Here's an overview of this research study.

| Purpose of Research Study | The purpose of this study is to determine if a food pantry network's transition to online ordering influences food security status among low-income adults and if there are differences by age group. We are asking you to take part in this study because you are at least 18 years old. |
|---|---|
| Key Information | The study will last about 18 months. Participation in this study involves a baseline visit and a follow-up data collection period/visit over the course of up to 8 months. You will be asked to complete surveys and have the food items you select at the food pantry documented. |
| Potential Risks | The most common risk is frustration from answering survey questions. |

Intervention Arm 

| Potential Benefits | You will not personally benefit from being in this study. Information from this study may provide evidence to be used in evaluating the effect of food pantries' transitioning to online ordering on clients' food selection. |
|---|---|
| Alternatives to Participation | Taking part in this study is voluntary. You can continue using the food pantry now and in the future without being in this study. |

More information about these topics can be found in the pages that follow. If you are interested in learning more, please review the rest of this document.

#### 2. About volunteering for this research study

Your participation is voluntary which means you can choose whether or not you want to take part in this study. People who agree to take part in research studies are called "subjects" or "research subjects". These words are used throughout this form. Before you can make your decision, you will need to know what the study is about, the possible risks and benefits of being in this study, and what you will have to do in this study. You may also decide to discuss this study and this form with your family or friends. If you have any questions about this study or this form, please ask us. If you decide to take part in this study, you must be asked to provide verbal consent. We will give you a copy of this form to keep.

## 3. What is the purpose of this study?

The purpose of this study is to see if a choice-based food pantry network's transition to online ordering influences food security status among low-income adults and if there are differences by age group.

# 4. How long will I be in the study? How many other people will be in the study?

Participation in this study involves a baseline visit and a follow-up data collection period/visit over the course of up to 8 months. The baseline visit will be in person at the food pantry. The follow up data collection/visit will take place virtually. The total duration for both of the data collection periods/visits will be 30-50 minutes. We anticipate up to 386 people will be in this study.

## 5. What will I be asked to do in the study?

If you choose to take part in the study, we will ask you to provide verbal consent first.

- During the Baseline period/visit:
  - This will take place in-person at the food pantry.
  - You will be asked to complete an in-person survey about your food and nutrition security, diet behaviors, and frequency of food pantry visits. This will take about 10 minutes. Survey responses will be collected using Qualtrics.

Intervention Arm 

- You will be given a card with an appointment time of your choosing that falls within the follow-up period. The card will include the phone number for a study team member in case you need to reschedule.
- A member of the study team will record the food items you select. This will take about 5 minutes

#### During the Follow-up period/visit:

- o We will send you follow-up reminders by email and/or text, based on your preference.
- You will be asked to complete a survey by phone about your food and nutrition security, diet behaviors, and frequency of food pantry visits. This will take about 10 minutes.
- You will be asked to give us permission to use data on your food item selections that will be gathered from the food pantry online ordering system. This data will be provided to the research team by the Met Council Kosher Food Pantry Network.

You are free to skip any questions you prefer not to answer. Any identifiable information collected and/or used for the purposes of this research will not be used or distributed for future research studies.

#### 6. What are the possible risks or discomforts?

There is a risk of breach of confidentiality. We will collect names, phone numbers, email addresses, and mailing addresses in a secure REDCap form only to facilitate data collection and gift card distribution in the follow-up period/visit. The REDCap data will not be linked to your Qualtrics survey responses.

The research team may need to communicate with you about information relevant to this research study. The research team will usually contact you for these purposes by phone, but if you have given the Researchers your email address and mobile/cell phone number and permission to send a text message, the research team may contact you that way. When the research team sends email messages that include identifiable health information, they will use encrypted messaging (e.g. SendSafe). When the research team uses texting over mobile/cell phones there is no way to encrypt the message. This means that the information you send or receive by text message is unencrypted and could be intercepted or viewed by an unintended recipient, or by your mobile/cell phone provider or carrier. Therefore, text messages carry security and privacy risks.

Below are some important points about texting in this research study:

- Text messages are not encrypted, and therefore are unsecure and may result in a breach of your confidentiality.
- You will be responsible for all fees charged by your carrier's service plan for text messaging. This
  research study and NYU Langone Health will not cover the cost related to any increased charges,
  data usage against plan limits or changes to data fees from the research texts
- Text messages will only be read during regular business hours. However, if you have a scheduled visit outside of business hours, you may receive a text in relation to this visit outside of regular business hours.

Intervention Arm 

- Text messaging should not be used in case of an emergency. If you experience an emergency, call 911 or go to the nearest hospital emergency department.
- You may decide to not send or receive text messages with staff associated with this research study at any time. You can do this in person or by sending the research number a text message that says "Stop Research Text."
- Your agreement applies to this research study only. Agreeing to other texts from NYU Langone
  Health for example appointment reminders, is a separate process. Opting out of other texts from
  NYU Langone Health is a separate process as well.

| he study. | | | | · · |
|---|---|---|---|---|
| | YES, I agree to receive texts from this resear | arch group. Initial | nere: | Cell phone |
| | number: | | | |

**NO**, I do not agree to receive texts from this research group. Initial here:

Please make sure to keep the research team updated if your mobile/cell phone number changes during

#### 7. What if new information becomes available?

During the course of this study we may find more information that could be important to you. This includes information that might cause you to change your mind about being in the study. We will notify you as soon as possible if such information becomes available.

## 8. What are the possible benefits of the study?

There are no direct benefits to you from being in this study. Information from this study may provide evidence to be used in evaluating the effect of food pantries' transitioning to online ordering on clients' food selection.

## 9. What other choices do I have if I do not participate?

Participating in this study is voluntary. Should you choose not to participate, you can continue using the food pantry without being in this research study. Your decision will not affect your ability to use the food pantry now or in the future.

## 10. Will I be paid for being in this study?

You will be paid by gift card for being in this study. If you chose to leave or are withdrawn from the study for any reason before finishing the entire study, you will be paid for each completed data collection period/visit.

You will be paid \$30 for completing the baseline data collection period/visit. You will be paid an additional \$50 for completing the follow-up data collection period/visit. If you complete both data collection periods/visits, you will be paid a total of \$80. After the baseline data collection visit, you will receive a

Intervention Arm 

physical gift card. Since the follow-up data collection visit will be virtual, you will receive either an e-gift card in your email or a physical gift card in the mail, depending on your preference.

You are required to track all payments made to you by NYU Langone Health for your participation in any research for this calendar year. You must let us know immediately if/when the total research payments presently equal or is likely to exceed \$600.00 total (not including travel reimbursements) for this calendar year. If your total payments (for one or more studies) reach \$600.00, please advise Dr. Rummo at Pasquale.Rummo@nyulangone.org.

In order to receive payments for your participation in research, you may need to provide your Social Security number. This is because NYU Langone Health is required to report to the IRS any amounts that are paid to research participants that are equal to or greater than \$600.00, and you may be taxed on these research payments above \$600.00. If you will receive payments in any amount by a check, you will need to provide your Social Security number or Alien Registration number and will be asked to complete a IRS W-9. If you do not have either of these numbers or are not willing to complete the W-9, you may be in the study but will not receive any payment.

#### 11. Will I have to pay for anything?

The study team may communicate with you by text if you agree to that method of communication. You will be responsible for all fees charged by your carrier's service plan for text messaging. This research study and NYU Langone Health will not cover the cost related to any increased charges, data usage against plan limits or changes to data fees from the research texts.

## 12. What happens if I am injured from being in the study?

We do not anticipate any risks of physical injuries as a result of being in this study. There are no plans for the NYU Langone Health to pay you or give you other compensation for injuries. You do not give up your legal rights by signing this form.

## 13. When is the study over? Can I leave the Study before it ends?

The overall study will last about 18 months. This study may be stopped or your participation ended at any time without your consent because:

- The principal investigator feels it is necessary for your safety. Such an action would not require your consent, but you will be informed if such a decision is made and the reason for this decision.
- You have not followed study instructions.
- The study sponsor, the principal investigator or other body responsible for monitoring the safety of the study has decided to stop the study.

If you decide to participate, you are free to leave the study at anytime. Leaving the study will not interfere with your ability to use the food pantry now or in the future.

## 14. How will you protect my confidentiality?

Intervention Arm 

We will collect your name, phone number, email address, and mailing addresses in a secure REDCap form for the purpose of facilitating the follow-up data collection, which will be conducted virtually, and to distribute gift cards. The REDCap data will not be linked to your Qualtrics survey responses.

#### **Certificate of Confidentiality**

To help us further protect your confidentiality, this research is covered by a Certificate of Confidentiality from the National Institutes of Health (NIH). The NIH has issued a Certificate of Confidentiality for this research. This adds special protection for the research information (data, documents, or biospecimens) that may identify you.

Research information protected by this Certificate of Confidentiality cannot be disclosed to anyone else who is not connected with the research, without your consent. With this Certificate of Confidentiality, the researchers may not disclose or use research information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence, for example, if there is a court subpoena, without your consent. However, disclosure, without your consent, is still necessary if there is a federal, state, or local law that requires disclosure (such as to report child abuse or communicable diseases).

The Certificate of Confidentiality cannot be used to refuse a request for information from appropriate government agencies responsible for project oversight.

The Certificate of Confidentiality does not prevent you from releasing information about yourself and your involvement in this research. Federal regulations may also allow for the use or sharing of information for other scientific research.

#### What information may be used or shared with others in connection with this study?

All information in your research record for this study may be used and shared with those individuals listed in this section.

#### Who may use and share information in connection with this study?

The following individuals may use, share, or receive your information for this research study:

- The research team, including the Principal Investigator, study coordinators, and personnel responsible for the support or oversight of the study
- The study sponsor: National Institute on Aging (NIA)
- Governmental agencies responsible for research oversight (e.g., the U.S. Food and Drug Administration or FDA).

## 15. The Institutional Review Board (IRB) and how it protects you

The IRB reviews all human research studies – including this study. The IRB follows Federal Government rules and guidelines designed to protect the rights and welfare of the people taking part in the research studies. The IRB also reviews research to make sure the risks for all studies are as small as possible. The NYU Langone Health IRB Office number is 212-263-4110. The NYU Langone Health IRB is made up of doctors, nurses, non-scientists, and people from the Community.

Intervention Arm 

# 16. Who can I call with questions, or if I'm concerned about my rights as a research subject?

If you have questions, concerns or complaints regarding your participation in this research study or if you have any questions about your rights as a research subject, you should speak with the Principal Investigator listed on top of the page 1 of this consent form. If a member of the research team cannot be reached or you want to talk to someone other than those working on the study, you may contact the NYU Langone Health IRB at 212-263-4110.

Do you have any questions? When you provide consent verbally, you are agreeing to take part in this research study as described to you. This means that you have read this form, your questions have been answered, and you have decided to participate in this study. Do you provide consent to take part in this study?